CLINICAL TRIAL: NCT03406052
Title: An Innovative Smartphone-enabled Health Coaching Intervention for Youth Diagnosed With Major Depressive Disorders
Brief Title: Smartphone-enabled Health Coaching Intervention for Youth Diagnosed With Major Depressive Disorders
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: New funding required
Sponsor: York University (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Yorku; 2016-115 (Other: Centre for Addiction and Mental Health); 2017-154 (Other Grant/Funding Number: Federal Development Program - S. Ontario)
Record Dates: First submitted 2017-12-04; First posted 2018-01-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Disorder, Major Depressive
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Psychiatrists providing psychiatric care will be blinded to the group allocation of subjects under their treatment. One outcome assessor (who will conduct the 24-item Hamilton Rating Scale for Depression (HRSD-24) will be blinded. Investigators will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-Assisted MB-CBT (Experimental): Online intervention accessed through smartphone or online accessed computer comprised of Mindfulness-Based Cognitive Behaviour content
  Interventions: Behavioral: Smartphone-Assisted MB-CBT
- Control (No Intervention): Standard psychiatric care

INTERVENTIONS:
Behavioral: Smartphone-Assisted MB-CBT — Experimental subjects will receive a mindfulness-based CBT online software program workbook (in collaboration with Nex J Systems, Inc.) accessible online. Exposure to and interaction with the online workbook is combined with health coaching (duration of 24 total hours) primarily delivered in phone and software interactions. In addition, each participant will be given a Fitbit-HR Charge, a wearable bracelet that assesses physical steps and 24 hour heart rate in 5 second (averaged) durations (with related access to software that permits daily tracking).
  Arms: Smartphone-Assisted MB-CBT

SUMMARY:
Randomized controlled trial (RCT) comparing youth diagnosed with major depressive disorder treated with online mindfulness-based cognitive behavioural therapy vs. standard psychiatric care (as wait-list controls). Eligible subjects will be recruited from the wait-lists of the Centre for Addiction and Mental Health. N = 168 subjects will consist of youth from First Nations background (18-30 yrs) and youth from all other ethnic backgrounds stratified to two intervention groups and two wait-list control groups consisting of 50% First Nations youth and 50% youth of all other ethnic backgrounds.

DETAILED DESCRIPTION:
A high proportion (70%) of mental health problems appear before 25 yrs. and can become become long-standing, significant disorders that impair all life domains. Early signs of disorder left untreated is an acute problem for Canadian youth as 15-25 yrs is the most likely age-strata for diagnosable psychiatric disorders, substance dependencies and suicide. Progress in youth treatments that engage the tendencies of youth to respond to online internet contact are likely to be especially strategic.

In this randomized controlled trial (RCT) diagnosed depressed youth are treated with online mindfulness-based cognitive behavioural therapy (MB-CBT) and standard psychiatric care or just standard psychiatric care (as wait-list controls). Eligible subjects will be recruited from the wait-lists of the Centre for Addiction and Mental Health (CAMH), and from community-based practices and clinics proximal to CAMH. The consented 168 subjects will be from First Nations background (18-30 yrs) and from all other ethnic backgrounds, stratified into two intervention groups and two wait-list control groups.

Primary outcome is self reported depression using the Beck Depression Inventory II while secondary outcomes include self reported anxiety (Beck Anxiety Inventory), depression (Quick Inventory of Depressive Symptomatology, 24-item Hamilton Rating Scale for Depression (HRSD-24)), pain (Brief Pain Inventory) mindfulness (Five-Facet Mindfulness Questionnaire) and intervention costs.

If hypotheses are confirmed that youth can be effectively treated with online MB-CBT at reduced costs, effective treatment can be delivered to greater numbers with less geographic restriction.

ELIGIBILITY:
Inclusion Criteria

* 18-30 yrs
* First Nations background or other ethnicity
* BDI-II at mild-moderate levels (i.e., BDI-II score ≥ 14 and < 29 )
* diagnosis of major depressive disorder
* fluent in english
* diagnosis by a CAMH physician and diagnosis confirmed by a MINI International Neuropsychiatric Interview

Exclusion Criteria

* < 18 yrs and > 30 yrs
* BDI-II in severe range ≥ 29 or < 14
* does not qualify for diagnosis of major depressive disorder or diagnosis not confirmed by MINI International Neuropsychiatric Interview

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory II | Baseline, 3 months, 6 months
  Change from baseline self report of symptoms of depression

SECONDARY OUTCOMES:
Beck Anxiety Scale | Baseline, 3 months, 6 months
  Change from baseline self report of anxiety symptoms
Quick Inventory of Depressive Symptomatology | Baseline, 3 months, 6 months
  Change from baseline self report of symptoms of depression
Hamilton Depression Rating Scale (HRDS-24) | Baseline, 3 months, 6 months
  Change from baseline interview and interviewer rating of symptoms of depression
Five-Facet Mindfulness Questionnaire | Baseline, 3 months, 6 months
  Change from baseline self report of mindfulness experience
Brief Pain Inventory | Baseline, 3 months, 6 months
  Change from baseline self report of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Ritvo, PhD, Principal Investigator — York University
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guglietti CL, Daskalakis ZJ, Radhu N, Fitzgerald PB, Ritvo P. Meditation-related increases in GABAB modulated cortical inhibition. Brain Stimul. 2013 May;6(3):397-402. doi: 10.1016/j.brs.2012.08.005. Epub 2012 Sep 7. PMID 23022436
- [Result] Radhu N, Daskalakis ZJ, Guglietti CL, Farzan F, Barr MS, Arpin-Cribbie CA, Fitzgerald PB, Ritvo P. Cognitive behavioral therapy-related increases in cortical inhibition in problematic perfectionists. Brain Stimul. 2012 Jan;5(1):44-54. doi: 10.1016/j.brs.2011.01.006. Epub 2011 Feb 5. PMID 22037137
- [Result] Wayne N, Perez DF, Kaplan DM, Ritvo P. Health Coaching Reduces HbA1c in Type 2 Diabetic Patients From a Lower-Socioeconomic Status Community: A Randomized Controlled Trial. J Med Internet Res. 2015 Oct 5;17(10):e224. doi: 10.2196/jmir.4871. PMID 26441467
- [Result] Azam MA, Katz J, Fashler SR, Changoor T, Azargive S, Ritvo P. Heart rate variability is enhanced in controls but not maladaptive perfectionists during brief mindfulness meditation following stress-induction: A stratified-randomized trial. Int J Psychophysiol. 2015 Oct;98(1):27-34. doi: 10.1016/j.ijpsycho.2015.06.005. Epub 2015 Jun 25. PMID 26116778
- [Result] Arpin-Cribbie C, Irvine J, Ritvo P. Web-based cognitive-behavioral therapy for perfectionism: a randomized controlled trial. Psychother Res. 2012;22(2):194-207. doi: 10.1080/10503307.2011.637242. Epub 2011 Nov 28. PMID 22122217
- [Result] Azam MA, Katz J, Mohabir V, Ritvo P. Individuals with tension and migraine headaches exhibit increased heart rate variability during post-stress mindfulness meditation practice but a decrease during a post-stress control condition - A randomized, controlled experiment. Int J Psychophysiol. 2016 Dec;110:66-74. doi: 10.1016/j.ijpsycho.2016.10.011. Epub 2016 Oct 18. PMID 27769879
- [Result] Pludwinski S, Ahmad F, Wayne N, Ritvo P. Participant experiences in a smartphone-based health coaching intervention for type 2 diabetes: A qualitative inquiry. J Telemed Telecare. 2016 Apr;22(3):172-8. doi: 10.1177/1357633X15595178. Epub 2015 Jul 21. PMID 26199275
- [Result] Croarkin PE, Levinson AJ, Daskalakis ZJ. Evidence for GABAergic inhibitory deficits in major depressive disorder. Neurosci Biobehav Rev. 2011 Jan;35(3):818-25. doi: 10.1016/j.neubiorev.2010.10.002. Epub 2010 Oct 12. PMID 20946914
- [Result] Levinson AJ, Fitzgerald PB, Favalli G, Blumberger DM, Daigle M, Daskalakis ZJ. Evidence of cortical inhibitory deficits in major depressive disorder. Biol Psychiatry. 2010 Mar 1;67(5):458-64. doi: 10.1016/j.biopsych.2009.09.025. Epub 2009 Nov 17. PMID 19922906
- [Derived] Walters C, Gratzer D, Dang K, Laposa J, Knyahnytska Y, Ortiz A, Gonzalez-Torres C, Moore LP, Chen S, Ma C, Daskalakis Z, Ritvo P. The Use of Text Messaging as an Adjunct to Internet-Based Cognitive Behavioral Therapy for Major Depressive Disorder in Youth: Secondary Analysis. JMIR Form Res. 2024 May 31;8:e40275. doi: 10.2196/40275. PMID 38820586
- [Derived] Dang K, Ritvo P, Katz J, Gratzer D, Knyahnytska Y, Ortiz A, Walters C, Attia M, Gonzalez-Torres C, Lustig A, Daskalakis Z. The Role of Daily Steps in the Treatment of Major Depressive Disorder: Secondary Analysis of a Randomized Controlled Trial of a 6-Month Internet-Based, Mindfulness-Based Cognitive Behavioral Therapy Intervention for Youth. Interact J Med Res. 2023 Dec 8;12:e46419. doi: 10.2196/46419. PMID 38064262
- [Derived] Ritvo P, Knyahnytska Y, Pirbaglou M, Wang W, Tomlinson G, Zhao H, Linklater R, Bai S, Kirk M, Katz J, Harber L, Daskalakis Z. Online Mindfulness-Based Cognitive Behavioral Therapy Intervention for Youth With Major Depressive Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 10;23(3):e24380. doi: 10.2196/24380. PMID 33688840